CLINICAL TRIAL: NCT04818632
Title: A Phase 1 Dose Escalation and Expansion Study of AZD9833 Alone or in Combination With Palbociclib or Everolimus in Chinese Patients With Oestrogen Receptor Positive (ER+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Metastatic Breast Cancer (mBC)
Brief Title: AZD9833 China PK Study
Acronym: AZD9833
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8530C00007
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2023-10

CONDITIONS: ER+, HER2-, Metastatic Breast Cancer
Keywords: Breast Cancer; Open-label; Phase 1; Safety; Tolerability; Pharmacokinetics; ER Positive; HER2 Negative; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833; palbociclib; Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AZD9833 monotherapy dose escalation (Experimental)
  Interventions: Drug: AZD9833
- AZD9833 monotherapy dose expansion (Experimental)
  Interventions: Drug: AZD9833
- AZD9833 with palbociclib dose expansion (Experimental)
  Interventions: Drug: AZD9833 with palbociclib
- AZD9833 with everolimus dose expansion (Experimental)
  Interventions: Drug: AZD9833 with everolimus

INTERVENTIONS:
Drug: AZD9833 — Part A: AZD9833 monotherapy dose escalation.
  Arms: AZD9833 monotherapy dose escalation
Drug: AZD9833 — Part B: AZD9833 monotherapy dose expansion
  Arms: AZD9833 monotherapy dose expansion
Drug: AZD9833 with palbociclib — Part B: AZD9833 with palbociclib dose expansion
  Arms: AZD9833 with palbociclib dose expansion
Drug: AZD9833 with everolimus — Part B: AZD9833 with everolimus dose expansion
  Arms: AZD9833 with everolimus dose expansion

SUMMARY:
A Phase 1 Dose Escalation and Expansion Study of AZD9833 Alone or in Combination in Chinese patients with ER Positive, HER2 Negative, Metastatic Breast Cancer

DETAILED DESCRIPTION:
This study is designed to investigate and characterize the safety, tolerability and PK of AZD9833 monotherapy (Part A, Part B-cohort 1) or in combination with palbociclib (optional Part B cohort 2) or everolimus (optional Part B cohort 3) and to explore the preliminary anti-tumour activity in Chinese patients

ELIGIBILITY:
Inclusion Criteria:

1. Any menopausal status:

   1. Pre-menopausal women must have commenced treatment with an LHRH agonist at least 4 weeks prior to the start of study intervention and must be willing to continue to receive LHRH agonist therapy for the duration of the study.
   2. Post-menopausal defined according to standard criteria in the protocol.
2. Histological or cytological confirmation of adenocarcinoma of the breast.
3. Documented positive ER status and HER2 negative status of primary or metastatic tumour tissue.
4. ECOG performance status 0 to 1.
5. Metastatic disease and radiological or objective evidence of progression on or after the last systemic therapy prior to the start of study intervention.
6. At least one lesion as per RECIST Version 1.1 that can be accurately assessed at baseline and is suitable for repeated assessment by CT, MRI, or plain X-ray or clinical examination.
7. Recurrence or progression on at least one line of endocrine therapy in the metastatic disease setting.
8. For Part A and Part B cohort 1, patients should be eligible for SERD monotherapy treatment.
9. For Part B Cohort 2, patients should be eligible for SERD treatment and CDK4/6 inhibitors, and prior treatment with CDK4/6 inhibitors is not permitted.
10. For Part B Cohort 3, patients should be eligible for SERD treatment and mTOR inhibitors, and prior treatment with mTOR inhibitors is not permitted.

Exclusion Criteria:

1. Previous treatment with AZD9833.
2. Presence of life-threatening metastatic visceral disease, uncontrolled CNS metastatic disease or life-threatening extensive hepatic involvement.
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, or infection requiring intravenous antibiotic therapy, which makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol.
4. Inadequate bone marrow reserve or organ function.
5. Any clinically important and symptomatic heart disease.
6. Any concurrent anti-cancer treatment.
7. Refractory nausea and vomiting, uncontrolled chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of AZD9833 (and palbociclib and everolimus).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pre-menopausal or Post-menopausal women
Enrollment: 28 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicity, as defined in the protocol. | Minimum observation period 28 days on treatment.
  Dose-limiting toxicity as described in the protocol that is not related to disease progression, intercurrent illness or concomitant medications and that, despite optimal therapeutic intervention, meets protocol-defined criteria of AZD9833 monotherapy. [part A only]
The number of subjects with treatment-related adverse events as assessed by CTCAE v5.0. | 6 months after the last patient recruited starts study intervention or 28 days after the final patient discontinues study intervention
  Data will include clinical observations, ECG parameters, clinical chemistry and haematology and vital signs assessed as the number of subjects with treatment-related adverse events assessed by CTCAE v5.0 of AZD9833 monotherapy.
Plasma AZD9833 concentrations and derived PK parameters. | At predefined intervals throughout the AZD9833 treatment period (approximately 16 weeks )
  To characterise the single- and multiple-dose PK of AZD9833 monotherapy.

SECONDARY OUTCOMES:
The number of subjects with treatment-related adverse events as assessed by CTCAE v5.0. | 6 months after the last patient recruited starts study intervention or 28 days after the final patient discontinues study intervention
  Data will include clinical observations, ECG parameters, clinical chemistry and haematology and vital signs assessed as the number of subjects with treatment-related adverse events assessed by CTCAE v5.0 of AZD9833 administered in combination with palbociclib or everolimus..
Plasma AZD9833 concentrations and derived PK parameters (for optional expansion cohorts Part B Cohorts 2 and 3 only). Everolimus (whole blood) concentrations and derived PK parameters (for optional expansion cohort Part B Cohort 3 only). | At predefined intervals throughout the AZD9833 treatment period (approximately 16 weeks )
  To characterise the single- and/or multiple-dose PK of AZD9833 administered in combination with palbociclib, and single- and/or multiple-dose PK of both AZD9833 and everolimus in combination.
Objective Response Rate | Week 8 and week 16 and week 24 and then every 12 weeks (week 36, 48, 60) until the end of the study (approximately 1 year)
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Duration of Response | Week 8 and week 16 and week 24 and then every 12 weeks (weeks 36, 48 and 60) until the end of the study (approximately 1 year)
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Clinical benefit rate at 24 weeks | Up to 24 weeks
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Percentage Change in Tumour Size | Week 8 and week 16 and week 24 and then every 12 weeks (weeks 36, 48 and 60) until the end of the study (approximately 1 year)
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Progression Free Survival | From start of treatment to disease progression/latest date of evaluable RECIST assessment (approximate 1 year)
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, Principal Investigator — Department of Breast Surgery, Fudan University Shanghai Cancer Center; Jian Zhang, Principal Investigator — Department of Medical Oncology, Fudan University Shanghai Cancer Center
Locations (4):
- China (4):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Shanghai
  - Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: AstraZenecaClinicaltrials.com — https://www.astrazenecaclinicaltrials.com/study/D8530C00007/